CLINICAL TRIAL: NCT02241850
Title: Assessment of Genetic Polymorphisms Affecting Effect of High Intensity Training in Korean Healthy Volunteers
Brief Title: Genetic Polymorphisms Affecting Effect of High Intensity Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Sung-Vin Yim, M.D., Ph.D., Kyunghee University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DW-HIT01
Record Dates: First submitted 2014-09-01; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: High Intensity Training; Genetic Polymorphisms; Genome Wide association study; Single Nucleotide Polymorphism genotype; Subjects
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High intensity training (Other): 9 weeks of supervised training
  Interventions: Other: High intensity training

INTERVENTIONS:
Other: High intensity training — 9 weeks of supervised high intensity training

SUMMARY:
The objective of the study is to investigate the effect of high intensity training on maximal oxygen uptake according to the genetic polymorphisms in healthy Korean volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 to 60, healthy male subjects (at screening)
* Volunteer who totally understands the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Volunteer who has past or present history of any diseases following below; liver including hepatitis virus carrier, kidney, Neurology, immunology, pulmonary, endocrine, hematooncology, cardiology, mental disorder
* Subject who already participated in other trials in 30 days
* Subject who had whole blood donation in 2 months, or component blood donation in 1 months or transfusion
* Subject who smokes an average of 20 cigarettes/day or drink > 5 cups of coffee

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change of maximal oxygen uptake | Baseline and after 6, 9 weeks of training

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Vin Yim, MD, PhD, Principal Investigator — Kyung Hee University Hospital

REFERENCES:
- [Derived] Yoo J, Kim BH, Kim SH, Kim Y, Yim SV. Genetic polymorphisms to predict gains in maximal O2 uptake and knee peak torque after a high intensity training program in humans. Eur J Appl Physiol. 2016 May;116(5):947-57. doi: 10.1007/s00421-016-3353-7. Epub 2016 Mar 21. PMID 27001664